CLINICAL TRIAL: NCT00989222
Title: Volar Plating or External Fixation of Dorsally Displaced Fractures of the Distal Radius? A Prospective Randomized Study
Brief Title: Volar Plating or External Fixation of Dorsally Displaced Fractures of the Distal Radius?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Responsible Party: Dr Maria Wilcke, Division of Orthopaedics, Karolinska Institutet, Department of Clinical Sciences, Danderyd Hospital, Stockholm, Sweden.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005/4:8
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2009-10-05 (Estimated); Status verified 2009-10

CONDITIONS: Radius Fractures
Keywords: Distal radius fractures; Fractures of the distal radius; Volar plate; External fixation
MeSH Terms: conditions — Radius Fractures; Wrist Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volar locked plate (Other): Open reduction and fixation of a unstable dorsally displaced fracture of the distal radius with a volar locked plate
  Interventions: Procedure: Internal fixation with a volar locked plate
- External fixation (Other): Fixation of an unstable dorsally displaced fracture of the distal radius with bridging external fixation
  Interventions: Procedure: closed reduction and external fixation

INTERVENTIONS:
Procedure: closed reduction and external fixation — Fixation of an unstable dorsally displaced fracture of the distal radius with bridging external fixation
  Other Names: External fixation: Hoffman compact
  Arms: External fixation
Procedure: Internal fixation with a volar locked plate — Open reduction and fixation of a unstable dorsally displaced fracture of the distal radius with a volar locked plate
  Other Names: Volar locked plate brand: Königsee by Swemac
  Arms: Volar locked plate

SUMMARY:
Promising results have been reported after volar locked plating of unstable dorsally displaced fractures of the distal radius. It offers stable fixation and early mobilization. The investigators' aim is to test if volar locked plating results in better patient-perceived, objective functional and radiological outcomes compared to the less invasive external fixation that has been the standard operation for decades.

ELIGIBILITY:
Inclusion Criteria:

* An acute unilateral Colles' fracture (AO class A and C1) with a dorsal angulation of more than 20 degrees or radial shortening of 4 mm or more, AND
* Patient aged 20-70 years with no previous fracture of either wrist.

Exclusion Criteria:

* Bilateral fractures,
* Other current injury to the upper extremities,
* Dementia, OR
* Severe comminution or too small distal fragment to allow plating.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
PRWE (patient rated wrist evaluation) score | 3,6 and 12 months

SECONDARY OUTCOMES:
Objective function (range of movement and grip strength) | 3,6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gustaf Neander, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Division of Orthopaedics, Karolinska Institutet, Department of Clinical Sciences, Danderyd Hospital, Stockholm, Sweden